CLINICAL TRIAL: NCT04737239
Title: Corticosteroid Injection Effectiveness in Carpel Tunnel Patients With Negative or Mild EMG
Brief Title: Corticosteroid Injection Effectiveness in Carpel Tunnel Patients With Negative or Mild EMG Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Other Study IDs: 14552
Record Dates: First submitted 2021-01-21; First posted 2021-02-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: corticosteroid injection; electromyography
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with CTS/Mild EMG
  Interventions: Other: Corticosteroid injections for CTS treatment
- Patient with CTS/Negative EMG
  Interventions: Other: Corticosteroid injections for CTS treatment

INTERVENTIONS:
Other: Corticosteroid injections for CTS treatment — Treatment of carpel tunnel syndrome with corticosteroid injections for EMG mild and EMG negative patients

SUMMARY:
Carpal Tunnel Syndrome (CTS) is the most common nerve entrapment syndrome worldwide. There are currently no studies examining the effectiveness of corticosteroid injections in patients with normal (negative) EMG studies. The purpose of this study is to gain a better understanding of the duration of symptom improvement post corticosteroid injection in patients with negative or mild EMG studies. The Boston Carpal Tunnel Questionnaire will be given to patients undergoing corticosteroid injections for the treatment of carpal tunnel syndrome to assess their response to the injection. Investigators will collect data retrospectively. The Boston Carpal Tunnel Questionnaire (BCTQ) is administered as per standard protocol to all patients with CTS who have a negative or mild EMG study. The BCTQ assesses the patient's self-reported symptom severity and functional status. Investigators will analyze this data with respect to demographics as well as numbness in the median n. distribution, nocturnal numbness, weakness/atrophy of the thenar musculature, Tinel's sign, Phalen's test, loss of 2-point discrimination, Quick-Dash score, and grip strength score.

The primary outcome will be the Boston Carpal Tunnel Questionnaire outcome score under the different EMG conditions.The secondary outcomes will be numbness in the median n. distribution, nocturnal numbness, weakness/atrophy of the thenar musculature, Tinel's sign, Phalen's test, loss of 2-point discrimination, QuickDash score, and grip strength score. Both outcomes will be examined in patients with negative or mild EMG readings. This information will allow orthopedic physicians to gain a better understanding of the duration of symptom improvement post-corticosteroid injection, allowing them to fine tune their treatment plans for CTS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who speak English
* Patients who are 18 years or older
* Patients who are clinically diagnosed with CTS
* Patients who have a negative or mild EMG study
* Patients who receive a corticosteroid injection after obtaining a negative or mild EMG study

Exclusion Criteria:

* Patients who do not speak English
* Patients who are younger than 18 years of age
* Patients who have experienced previous trauma to the wrist
* Patients who have had previous treatment for CTS including but not limited to corticosteroid injection or surgery
* Patients with a moderate or severe EMG study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients clinically diagnosed with CTS, have a negative or mild EMG study, and receive a corticosteroid injection at Henry Ford Health System Orthopedics.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Boston Carpel Tunnel Questionnaire | Dec 23 2020-Dec 22 2021
  Scaled 1-5, higher scores indicate worse outcomes

SECONDARY OUTCOMES:
Number of patients with numbness in the median n. distribution | Dec 23 2020-Dec 22 2021
  Positive test includes numbness in parts of palm, thumb, second and third finger, assessed by physician
Number of patients with weakness/atrophy of the thenar musculature | Dec 23 2020-Dec 22 2021
  Positive test includes weakness in grip or holding objects as described by participant, assessed by physician
Number of patients with positive Tinel's Sign | Dec 23 2020-Dec 22 2021
  Positive sign includes 'pins and needles' in parts of palm, thumb, second and third finger upon percussion of median nerve, assessed by physician
Number of patients with positive Phalen's Test | Dec 23 2020-Dec 22 2021
  Positive test includes pain in parts of palm, thumb, second and third finger associated with compression of the median nerve, assessed by physician
2-point discrimination Test | Dec 23 2020-Dec 22 2021
  Scaled 2-8mm, higher scores indicate worse outcomes
QuickDash score | Dec 23 2020-Dec 22 2021
  Scaled 1-100, higher scores indicate worse outcomes
Grip Strength score | Dec 23 2020-Dec 22 2021
  Scored in pounds(lbs), higher scores indicate better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Graham B, Regehr G, Naglie G, Wright JG. Development and validation of diagnostic criteria for carpal tunnel syndrome. J Hand Surg Am. 2006 Jul-Aug;31(6):919-24. PMID 16886290
- [Background] Visser LH, Ngo Q, Groeneweg SJ, Brekelmans G. Long term effect of local corticosteroid injection for carpal tunnel syndrome: a relation with electrodiagnostic severity. Clin Neurophysiol. 2012 Apr;123(4):838-41. doi: 10.1016/j.clinph.2011.08.022. Epub 2011 Oct 1. PMID 21962473